CLINICAL TRIAL: NCT00326742
Title: Validation in Humans of Genes Involved in Alcohol Drinking, Stress-Induced Alcohol Drinking and Relapse
Status: Completed | Type: Observational
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Other Study IDs: NGFN 2 01 GS 0475
Record Dates: First submitted 2006-05-16; First posted 2006-05-17 (Estimated); Last update posted 2007-05-10 (Estimated); Status verified 2007-05

CONDITIONS: Alcohol Drinking
Keywords: Alcoholism; Risk factors; Adolescence; Stress test; HPA system; Family adversity; Candidate genes; Cortisol; Adrenocorticotrophin
MeSH Terms: conditions — Alcohol Drinking; Alcoholism | interventions — Psychological Tests

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Behavioral: Trier Social Stress Test

SUMMARY:
Aim of the project is to validate and functionally characterize the combined impact of candidate genes and stress exposure on drinking in adolescents. Lifetime and recent stress experiences and drinking are recorded in a sample of healthy young adults who are genotyped for polymorphisms in candidate genes related to alcoholism. All participants undergo a standard laboratory psychosocial stress test. Our hypothesis is that specific genes can be identified which influence drinking by modulating stress response.

ELIGIBILITY:
Inclusion Criteria:

* All 18 or 19 year old participants of the Mannheim risk children study, i.e. a longitudinal birth cohort study that started in 1986 and had the inclusion criteria given below:
* Male and female singletons, firstborn to their mothers between February 1st, 1986 and February 28th, 1988, consecutively recruited from 2 obstetric and 4 children's hospitals of the Rhine-Neckar region, Germany.
* with no severe physical handicaps, obvious genetic defects, or metabolic diseases.
* with German-speaking Caucasian parents.
* Falling into one of 3 predefined groups with absent, moderate or high pre- and perinatal risk, operationalized by low gestational age at birth, low birth weight, and severity of the following: Preterm labor, EPH-gestosis, perinatal asphyxia, seizures, respiratory distress syndrome, perinatal sepsis.
* Falling into one of 3 predefined groups with absent, moderate or high psychosocial risk, operationalized by a family risk index measuring the presence of 11 adverse family factors covering characteristics of the parents (e.g., psychiatric disorders), the partnership (e.g., disharmony), and the family environment (e.g., overcrowding)during a period of one year prior to birth.

Exclusion Criteria:

* Intelligence quotient or motor quotient below 70, or presence of severe neurological disorder such as infantile cerebral palsy, at age 15.
* Women with known pregnancy.
* Any physical of psychiatric disease requiring treatment
* Incapable to give informed consent or to answer questionnaires in writing
* Recent use of illegal drugs

Ages: 18 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 281 (Actual)
Dates: Start 2005-07; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl F Mann, Prof, Principal Investigator — Central Institute of Mental Health, Mannheim
Locations (1):
- Department of Addictive Behavior und Addiction Medicine, Central Institute of Mental Health, Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Zimmermann U, Spring K, Kunz-Ebrecht SR, Uhr M, Wittchen HU, Holsboer F. Effect of ethanol on hypothalamic-pituitary-adrenal system response to psychosocial stress in sons of alcohol-dependent fathers. Neuropsychopharmacology. 2004 Jun;29(6):1156-65. doi: 10.1038/sj.npp.1300395. PMID 15100697
- [Background] Laucht M, Esser G, Schmidt MH. Developmental outcome of infants born with biological and psychosocial risks. J Child Psychol Psychiatry. 1997 Oct;38(7):843-53. doi: 10.1111/j.1469-7610.1997.tb01602.x. PMID 9363583
- See also: Homepage of the Department conducting the study — http://www.zi-mannheim.de